CLINICAL TRIAL: NCT02365103
Title: Investigation Into the Inhibitory Effects of Tea Consumption on Iron Bioavailability in a Cohort of Healthy United Kingdom (UK) Women, Using a Stable Iron Isotope
Brief Title: Tea Consumption and Iron Bioavailability in Women Using a Stable Isotope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14/NW/0310 S-LS17042014
Record Dates: First submitted 2015-02-04; First posted 2015-02-18 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Anemia, Iron-Deficiency; Iron, Bioavailability; Hepcidins; Intestinal, Absorption; Isotope Labeling, Stable
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Water; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test meal I (given with water) (Other): Test meal with water
  Interventions: Other: Test meal I (given with water)
- Test meal II (simultaneously with tea) (Other): Test meal with tea (simultaneously)
  Interventions: Other: Test meal II (simultaneously with tea)
- Test meal III (1 hour after test meal) (Other): Test Meal with tea given 1 hour after test meal
  Interventions: Other: Test meal III (1 hour after test meal)
- Reference Iron Dose (Other): Reference iron dose administered
  Interventions: Other: Reference iron dose

INTERVENTIONS:
Other: Test meal I (given with water) — 4 mg of the iron stable isotope, in a form of ferrous sulphate solution, extrinsically labelled in the test meal administered in the study, enrichment in the system will take approximately 14 days post dosing
  Arms: Test meal I (given with water)
Other: Test meal II (simultaneously with tea) — 4 mg of the iron stable isotope, in a form of ferrous sulphate solution, extrinsically labelled in the test meal administered in the study, enrichment in the system will take approximately 14 days post dosing
  Arms: Test meal II (simultaneously with tea)
Other: Test meal III (1 hour after test meal) — 4 mg of the iron stable isotope, in a form of ferrous sulphate solution, extrinsically labelled in the test meal administered in the study, enrichment in the system will take approximately 14 days post dosing
  Arms: Test meal III (1 hour after test meal)
Other: Reference iron dose — 3 mg of the iron stable isotope, in a form of ferrous sulphate solution, extrinsically labelled and administered in the study, enrichment in the system will take approximately 14 days post dosing
  Arms: Reference Iron Dose

SUMMARY:
The purpose of this study is to investigate the inhibition effect of tea consumption on non haem iron absorption with the use of an iron tracer. The study also aims to assess the effect of time variability of tea consumption on non haem iron absorption from a typical western breakfast.

DETAILED DESCRIPTION:
This is a non randomised controlled trial in 12 healthy participants over a period of 56 days. The study will investigate the inhibition effect of tea consumption on non haem iron absorption with the use of a stable iron isotope (Fe57) tracer. The study also aims to assess the effect of time variability of tea consumption on non haem iron absorption from a typical western breakfast.There is evidence of lower iron absorption when a meal is given with tea, compared to water. There is also evidence from previous studies that the inhibition effect is higher when tea is consumed simultaneously with a meal, compared to in between meals. However, there are limited number of human studies investigating iron absorption and time interval, particularly in the UK. The study aims to recruit 12 healthy participants. The test meals will be given together with black tea labelled with iron tracer, at various time intervals which includes together and after the meals. Test meal given with water will be used as a control. Blood samples will be collected 14 days post dosage for each of the meals. The study will take place at University of Chester, and participants will attend 5 clinics during the 56 day study. Prior to the start of study, participants will complete a 3 day food diary, where they will be given instructions by the researcher. In each clinic, weight and height will be measured, followed by a fasted blood sample and the administration of test meals.

PROJECT HYPOTHESES H1: There is a significant difference in non haem iron absorption from a typical western breakfast with tea consumption compared to without tea consumption H0:There is no significant difference in non haem iron absorption from a typical western breakfast with tea consumption compared to without tea consumption H1: Iron absorption will be lower when tea is consumed simultaneously with meals compared to when it is consumed in between meals H0: The iron absorption will not be lower when tea is consumed simultaneously with meals compared to when is consumed in between meals H1: There is an inverse correlation between tea consumption and iron status parameters H0: There is no inverse correlation between tea consumption and iron status parameters

There are several parameters which will be measured in this study. Height and weight will be measured using methods outlined in the Manual of Dietetic Practice using validated equipment (weighing scales and stadiometer). These will be measured by the student researcher at baseline and at each clinic (Clinic 1 to 5). Dietary intakes will be measured based on the data gathered in the 3 days food diary completed by the participants prior to Clinic 1 and 5. Additionally, blood samples will be taken by student researcher at each clinic. The analysis will be carried out in the Clinical Laboratories and Phlebotomy Room within the Department of Clinical Sciences and Nutrition (University of Chester), utilising the equipment and the clinical space where the participants will have to report during the administration of the meals with iron tracer. Test meals will be prepared in the food skills kitchen within the department. Analysis of blood samples will also be carried out in Clinical Sciences laboratories using relevant methodologies, including ELISA assays, bioanalysers and mass spectrometry. After the administration of meals labelled with iron tracers, all the blood samples will be stored at 80 Celsius in the laboratory until further analysis.

RECRUITMENT PROCESS The sampling will be carried out at the University of Chester. Posters/leaflets and letter/emails will be used as a medium of advertisement to the targeted group, especially to staff and students. The potential participants who require further information will be given participant information sheet which explains the procedure of the study.

STUDY PROCEDURE Clinic visits will take place between 0800 to 1000 (lasting for approximately 45 minutes) at the Clinical Sciences & Nutrition laboratory, University of Chester. 5 clinics are required, with a time interval of 14 days between clinics to allow the incorporation of the stable iron isotope (Fe57) tracer into the blood. During each clinic, participants will be given test meals labelled with iron tracer and tea, and no food or drink will be allowed for the next 3 to 4 hours. All the containers used to administer the test meals will be washed with ultrapure water to make sure complete consumption of both test meals and iron tracer. Participants will attend each clinic after an overnight fast (10 hours), and 30 ml blood samples (6 teaspoons) will be collected at each clinic. All the clinic details are given below.

Clinic 1 (Day 0): Participants will complete a screening questionnaire, followed by physical measurements of height and weight. If they satisfy the inclusion criteria, they will be invited to participate in the study and be asked to sign an informed consent form. Participants will be asked about their food consumption over the previous 24 hours and will be required to complete 3 day food diary to reflect habitual intake. Participants will be given an explanation on how to record the dietary intake. Height and weight will be measured, followed by a baseline blood sample. This will be followed by consumption of the control test meal.

Clinic 2 (Day 14): Measurement of height and weight followed by a baseline blood sample and 24 hour food recall will be carried out. This will be followed by consumption of the test meal II with tea given simultaneously with the test meal.

Clinic 3 (Day 28): Measurement of height and weight followed by a baseline blood sample and 24 hour food recall will be carried out . This will be followed by consumption of the test meal III with tea given 1 hour after the test meal.

Clinic 4 (Day 42): Measurement of height and weight followed by a baseline blood sample and 24 hour food recall will be carried out . This will be followed by consumption of reference dose iron.

Clinic 5(Day 56): Prior to the completion of the study, participants will be given another 3 day food diary which has to be completed before the clinic for another assessment of dietary intake. Measurement of height and weight followed by a final blood sample drawn to measure the incorporation of iron from the reference dose and 24 hour food recall.

DATA-PLAN

Sample size determination and justification :

Sample size was estimated using iron absorption data (mean ± S.D) from a study by Derman et al. (1977) in which they reported iron absorption (%) of 6.7 ± 6.2 when the test meals were administered with tea and 34.0 ± 23.0 when the test meals were administered without tea. With an effect size of 1.324, the total sample size required in the proposed study is 10. Taking into account a 20% drop out rate, the total sample size required to demonstrate a significant difference in iron absorption between consumption of meal with and without tea is 12 (Power = 0.95).

Data Analysis :

All statistical analyses will be conducted by the research student with International Business Machines (IBM)® Statistical Package for the Social Sciences (SPSS)® Statistic Data Editor Software (Version 21). Values for iron absorption and meal ratios will be expressed as geometric means and standard deviations. Iron absorption values (in percentage) will be logarithmically transformed for the purpose of analyses and will then be retransformed to recover the original units (Hurrell et al., 1999). Assuming that the data is normally distributed after performing normality test (Shapiro Wilks), paired student t tests will be conducted (i) to compare the iron absorption from each pair of meals and (ii) to obtain the absorption ratios in the test meals in relative to the reference dose without meal. Pearson's correlation test will be performed to investigate the relationship between tea drinking and iron status biomarkers. A nonparametric approach will be adopted if the data is not normally distributed for all analyses. Differences will be considered significant with a p value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* pre menopausal women;
* aged 19- 40 years;
* healthy;
* non- pregnant nor lactating.

Exclusion Criteria:

* history of gastrointestinal and metabolic disorders;
* have donated blood within past 6 months;
* regularly consuming nutritional supplements.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Iron absorption (%) measured by mass spectrometer | 14 days after each test meal
  Iron absorption is estimated based on the erythrocyte iron incorporation to the body system with the use of iron tracer after 14 days following administration of the test meals

SECONDARY OUTCOMES:
Serum ferritin measured by Biomerieux mini VIDAS | 1 year
  To assess the body iron storage
Hepcidin measured by enzyme-linked immunosorbent assay (ELISA) kit | 1 year
  To assess the mechanism involved in iron absorption
Full blood count measured by Beckman Coulter Counter | 1 year
  To assess the iron status
Zinc protoporphyrin (ZPP) measured by haemato-fluorimetry | 1 year
  To assess the iron status
Total binding iron capacity (TIBC) measured by enzyme-linked immunosorbent assay (ELISA) kit | 1 year
  To assess the total capacity of circulating transferrin bound to iron
Transferrin saturation measured by enzyme-linked immunosorbent assay (ELISA) kit | 1 year
  To assess the proportion of transferrin bound to iron
Transferrin receptor measured by enzyme-linked immunosorbent assay (ELISA) kit | 1 year
  To assess the severity of iron deficiency even in presence of inflammatory disorders
C- reactive protein measured by enzyme-linked immunosorbent assay (ELISA) kit | 1 year
  To assess levels of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Sohail Mushtaq, PhD, Principal Investigator — University of Chester
Locations (1):
- University of Chester, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The results are in the writing phase, and will be available in thesis form and possibly publication. It will be available in thesis form in 2017 and publication expected to be in 2018.

REFERENCES:
- [Background] Ahmad Fuzi SF, Koller D, Bruggraber S, Pereira DI, Dainty JR, Mushtaq S. A 1-h time interval between a meal containing iron and consumption of tea attenuates the inhibitory effects on iron absorption: a controlled trial in a cohort of healthy UK women using a stable iron isotope. Am J Clin Nutr. 2017 Dec;106(6):1413-1421. doi: 10.3945/ajcn.117.161364. Epub 2017 Oct 18. PMID 29046302